CLINICAL TRIAL: NCT02665494
Title: Biliary Cancer in Italy: a Study on Cholangiocarcinoma cAUSEs and Risk Factors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione del Piemonte per l'Oncologia (Other)
Responsible Party: Sponsor
Other Study IDs: BI-CAUSE
Record Dates: First submitted 2016-01-24; First posted 2016-01-27 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Multi-centric, observational, prospective study, designed for pts with diagnosis of all-stages cholangiocarcinoma, including rare and crossing-over histological types, and excluding gallbladder cancer and ampullary carcinoma.

DETAILED DESCRIPTION:
Patients will undergo basal blood sample exams regarding blood cell count, renal and liver function, tumor markers, inflammatory and metabolic state, along with a screening (and, if needed, a more in-depth laboratory analysis) for viral hepatitis infections. Information will be collected about radiological, clinical and pathological features of the neoplasm at time of diagnosis, as well, at a later time, about its natural history. A two-step data analysis will be performed: Task-1 analysis will define the risk factors landscape, Task-2 analysis will examine the influence of etiology on clinical outcomes. Anonymized data will be stored in a central database, kept at the Leading Centre.

ELIGIBILITY:
Inclusion Criteria:

* voluntary, written, dated and signed informed consent;
* age ≥ 18 years;
* histologically documented diagnosis of cholangiocarcinoma (including histological variants and mixed forms). Neoplasms under investigation do not include gallbladder cancer and ampullary carcinoma.

Exclusion Criteria:

* Dementia or altered mental status leading to inability to understand or render the informed consent.
* Patients who already underwent a systemic treatment (chemotherapy and/or targeted therapy) may be enrolled but will not be subject to data collection about BI-CAUSE - Study Protocol Version 1.0 Oct 18th, 2015 10 blood laboratory tests (with the exception of viral screening) and natural history, and will not be factored in the data analysis of prognostic factors. Performance status, life expectancy, tumour staging, tumour site (distal or hilar extrahepatic, intrahepatic), previous surgical resection, previous biliary stenting, previous radiotherapy are not part of inclusion/exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with diagnosis of all-stages cholangiocarcinoma, including rare and crossing-over histological types, and excluding gallbladder cancer and ampullary carcinoma
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
assessment the prevalence of a broad pool of medical or non-medical (e.g. life-style) conditions among Italian patients with cholangiocarcinoma, in order to evaluate their potential role as a risk factor | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Leone, MD, Principal Investigator — IRCCS Candiolo
Locations (12):
- Italy (12):
  - Istituto Tumori Giovanni Paolo II Bari - IRCCS, Bari, Bari
  - Ospedale Sant'Orsola Malpighi, Bologna, Bologna
  - Azienda Ospedaliera S.Croce e Carle Cuneo, Cuneo, Cuneo
  - Istituto Oncologico Veneto - IRCCS, Padua, Padova
  - Ospedale Santo Spirito di Pescara, Pescara, Pescara
  - Azienda Ospedaliero-Universitaria Pisana, Pisa, Pisa
  - Policlinico Universitario Campus Bio-Medico, Rome, Rome
  - Istituto Nazionale Tumori Regina Elena, Rome, Rome
  - Fondazione del Piemonte per l' Oncologia - IRCCS Candiolo, Candiolo, Torino
  - AOU Città della Salute e della Scienza di Torino - Ospedale Molinette, Turin, Turin
  - AO Ordine Mauriziano di Torino, Turin, Turin
  - Azienda Ospedaliero-Universitaria di Udine, Udine, Udine

IPD SHARING:
Plan to Share IPD: No